CLINICAL TRIAL: NCT07350161
Title: Implementation of a Caregiver-Report Suicide-Risk Screener in Children Under Age 8 in a Behavioral Health Center: A Pilot Study
Brief Title: Implementation of a Caregiver-Report Suicide-Risk Screener in Children Under Age 8 in a Behavioral Health Center
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 202501012; UL1TR002345 (NIH)
Record Dates: First submitted 2026-01-13; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Information Dissemination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- information group (Experimental): receives additional information about childhood SITBs
  Interventions: Other: SITB information
- no information group (No Intervention): does not receive additional information about childhood SITBs

INTERVENTIONS:
Other: SITB information — childhood SITB information
  Arms: information group

SUMMARY:
This project addresses the pressing need for tools to identify suicidal thoughts and behaviors in children aged 4-7. Although young children can experience STBs, current screening tools and guidelines often overlook this age group, partly due to challenges in directly assessing young children. The investigators developed a promising caregiver-report screener that identified at-risk children. This study will evaluate the screener's feasibility and effectiveness in clinical settings, gather feedback from clinicians and caregivers, and refine the screening process. The goal is to facilitate early intervention, improving mental health care and outcomes for young children.

DETAILED DESCRIPTION:
This project aims to evaluate the feasibility, acceptability, and efficacy of a caregiver-report suicide risk (STB) screening tool for children under age 8. Despite the rising rates of STBs in young children, tools for identifying at-risk individuals in this age group are limited, and significant resistance remains to screening children for STBs. Given the challenges in directly assessing young children and the lack of validated tools, the investigators developed a caregiver-report screener to detect early signs of STBs. Preliminary data indicate that this screener is both sensitive and specific, showing promise in identifying at-risk children. The proposed study will evaluate the implementation of this screener in a child behavioral health clinic, obtaining qualitative and quantitative feedback from both clinicians and caregivers to refine the screener and its integration into clinical workflows. Additionally, the investigators will assess how clinicians use the screener results in diagnostic and treatment planning. This study will provide critical insights into barriers and best practices for STB screening in young children, ultimately improving early identification and clinical care for at-risk youth.

ELIGIBILITY:
Inclusion Criteria:

* licensed mental health clinician (e.g., LPC, LMSW, LCSW, MD) in the Hermann Center
* provides care to children 4-7 years of age
* provides care through the Early Child Intervention, Early Psychiatric Care, or Trauma Response program
* must be currently seeing and/or accepting new patients

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-12-26 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Clinician report of SITB screen acceptability | From time of intervention until the follow-up interviews 3-4 months later.
  Interview data from clinicians will be qualitatively analyzed to identify patterns in feedback related to acceptability of the screen.

SECONDARY OUTCOMES:
Clinician report of hesitancies regarding use of SITB screen | From time of intervention until the follow-up interviews 3-4 months later.
  Interview data from clinicians will be qualitatively analyzed to identify patterns in feedback related to hesitancies with including the screen in the intake packet.
Clinicians' incorporation of SITB Screen in Child Treatment Plans | From time of intervention until the follow-up interviews 3-4 months later.
  Interview data from clinicians will be qualitatively analyzed to identify patterns in feedback related clinician's incorporation of the SITB screen results into their treatment plans.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
This is a very small pilot study with minimal resources for data sharing.